CLINICAL TRIAL: NCT06030869
Title: MyCustom:A Framework for Prospective and Master Protocol Trial of Precise Drug Treatment for Refractory Solid Tumors
Brief Title: MyCustom:Prospective Master Protocol Trial on Precision Medicine Treatment for Refractory Solid Tumors
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tianjin Medical University Second Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: MyCustom for Solid Tumors
Record Dates: First submitted 2023-09-02; First posted 2023-09-11 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2023-09

CONDITIONS: Refractory Solid Tumors; Next Generation Sequencing
Keywords: Precision medicine; NGS; Molecular Tumor Board(MTB)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Cohort-A: Patients with actionable targets: In the OncoKB(Precision Oncology Knowledge Base) database, the gene alteration has a variant of clinical evidence in this tumor or other tumor types and is considered to be an interventional variant. Cohort-A may include different observation subgroups. For example, substudy-A1: monotherapy/combination therapy for patients with A1-relative. Substudy-Ax: monotherapy/combination therapy for patients with Ax-relative.
- Cohort-B: Patients with potential actionable targets: In cohort-B, the gene alteration that MTB combines with clinical practice and literature reports that can match targeted therapy is considered to be potential actionable targets. Cohort-B also includes different observation subgroups and clinical trials may conduct in each subgroup. For example, substudy-B1(TP53 as driver gene), substudy-B2(RAS as driver gene), substudy-B3(MAP2K1 as driver gene), substudy-B4(PTEN Loss as driver gene), substudy-B5(11q13 co-amplification as driver genes), Substudy-B6(concomitant actionable alterations), substudy-B7(other driver genes). MTB-guided therapy was defined as having a clinical benefit if the PFS ratio between the longest PFS on MTB-guided therapy and the PFS on the last therapy before MTB-guided therapy was ≥1.3 (i.e., using patients as their own controls) for each substudy. To meet the primary objective, at least 35% of participants had to achieve a PF2S/PFS1 ≥ 1.3 in a sample population of 25 evaluable patients.
- Cohort-C: Patients with non-actionable targets: MTB combined with clinical practice and literature reports can not match the gene alteration of targeted therapy, which is considered as an irreversible gene alteration.

SUMMARY:
The MyCustom study is a investigator initiated trial(IIT), prospective real-world clinical research project, a genetic biomarker-driven "basket" (tissue-type agonistic) study. The target population covers a variety of solid advanced malignant tumors, including but not limited to patients with small cell lung, gastric, prostate, bladder cancer, head and neck squamous carcinoma or lacking effective treatment after standard treatment failure.

DETAILED DESCRIPTION:
The MyCustom study is a investigator initiated trial(IIT), prospective real-world clinical research project, a genetic biomarker-driven "basket" (tissue-type agonistic) study. The target population covers a variety of solid advanced malignant tumors, including but not limited to patients with small cell lung, gastric, prostate, bladder cancer, head and neck squamous carcinoma or lacking effective treatment after standard treatment failure.The overall goal is to develop a more effective research method to test new individualized treatment hypotheses.This study will provide comprehensive theoretical and practical support for individualized custom model in refractory solid tumors.Archival pathology laboratory samples from patients with treatment-refractory advanced solid cancer of any histologic type undergo Next Gene Sequencing(NGS) analysis.Fllowing obtain the raw data of the patient's gene sequencing, the data are analyzed by the auxiliary decision algorithm to obtain the prioritization results of the drugs matched by this patient.The results are subsequently reviewed by the Molecular Tumor Board (MTB), where eligible patients can be treated in treatment substudies.All patients who receive treatment with a drug available in the protocol will be followed for standard efficacy outcomes including clinical efficacy ,clinical safety and exploratory endpoints such as biomarkers for drug response, change in the tumor microenvironment. For some clinical studies, to meet the primary objective, at least 35% of participants had to achieve a PF2S/PFS1 ≥ 1.3 in a sample population of 25 evaluable patients. sample size was calculated using an exact single-stage design for phase II studies with a one-sided type I error of 5% and a power of 90% under the assumption that PF2S/PFS1≥ 1.3 in ≤10% of patients would be clinically irrelevant, while a success rate ≥ 35% would merit further investigation.

ELIGIBILITY:
Inclusion Criteria:

1. Adults(≥18 years of age)with pathologically confirmed advanced or metastatic solid cancer of any histological type, or an earlier diagnosis of cancer with a poor prognosis. Suffificient accessible tissue for molecular profifiling;
2. Patients receiving their last line of standard treatment or who have received and failed all standard anticancer therapy (if available) or are unsuitable for further standard anticancer therapy. Cancers with a poor prognosis or low expected response rate to standard treatment (as judged by the investigator on the basis of available evidence) may be screened with respect to an earlier line of treatment;
3. ECOG performance status of 0-4(Poor performance status caused by tumor diseases(3-4));
4. Willing and potentially able to comply with study requirements,including treatment, timing and nature of required assessments;
5. Signed, written informed consent to participate.

Exclusion Criteria:

1. Suitable for standard therapy;
2. Specific contraindications to exposure to the investigationalproducts;
3. Other comorbid conditions that may compromise assessing key outcomes or, in the judgement of the clinician, limit the ability of the patient to comply with the protocol;
4. Symptoms and uncontrolled central nervous system (CNS) involvement in a patient with a non-central cancer;
5. Pregnancy, lactation or inadequate contraception.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible patients have an advanced or metastatic solid tumor, multiple cancers(including but not limited to small cell lung cancer, gastric cancer, prostate cancer, bladder cancer, and head and neck squamous cell carcinoma) standard treatment options are no longer available or lack effective treatments.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
PFS2/PFS1(Progression Free Survival 2/Progression Free Survival 1) | 3 years
  The time to progression-free survival during the substudy (PFS2) exceeds the documented time to disease progression-free survival during the last treatment prior to substudy entry (PFS1) by at least 35% (ie, PFS2/PFS1≥1.3) or, if PFS1 is not evaluable, time to progressive disease exceeds 6 months.

SECONDARY OUTCOMES:
ORR(Objective Response Rate) | 3 years
  Evaluation of the best objective response rate (ORR) for each treatment according to RECIST 1.1. The best ORR is the best response reached during treatment according to RECIST 1.1 criteria.
OS(Overall Survival) | 3 years
  Evaluation of overall survival (OS) defined as the time between inclusion and death, whatever the cause is. Alive patients will be censored at their last known contact date.
Number of treatment related adverse events with grade 3 or greater severity by CTCAE 5.0 | 3 years
  Treatment related adverse events with grade 3 or greater severity by CTCAE 5.0.
Proportion of patients with actionable target | 3 years
  Number of patients with modifiable genomic variants.

CONTACTS AND LOCATIONS:
Overall Officials: Haitao Wang, Ph.D, Principal Investigator — Tianjin Medical University Second Hospital
Locations (1):
- Tianjin Medical University Second Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided